CLINICAL TRIAL: NCT01720654
Title: Expedited Partner Therapy as STI Control Among MSM in Peru
Brief Title: Expedited Partner Therapy for MSM in Peru
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Asociación Civil Impacta Salud y Educación, Peru (Other)
Responsible Party: Principal Investigator, Jesse Clark, Assistant Professor-in-Residence, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R21MH092232 (NIH); IMP-478-2012 (Other: Instituto Nacional de Salud del Peru); R21MH092232 (NIH)
Record Dates: First submitted 2012-10-29; First posted 2012-11-02 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Gonorrhea; Chlamydia
Keywords: Expedited Partner Therapy; MSM; Peru; Gonorrhea; Chlamydia
MeSH Terms: conditions — Gonorrhea; Chlamydia Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Standardized partner notification counseling.
- EPT (Experimental): Standardized partner notification counseling and provision of 5 partner treatment (EPT) packets.
  Interventions: Behavioral: EPT

INTERVENTIONS:
Behavioral: EPT — Standardized partner notification counseling and provision of 5 partner treatment packets containing: Printed information on signs, symptoms, diagnosis, and treatment of gonorrhea and chlamydia as well as information on local testing/treatment resources; 400 mg Cefixime and 1g Azithromycin.
  Arms: EPT

SUMMARY:
Expedited Partner Therapy (EPT) has been shown to reduce rates of persistent or recurrent gonorrhea and chlamydia infection in heterosexual patients, but has not been evaluated for use among men who have sex with men (MSM). CDC guidelines support the use of EPT for partner management with heterosexual patients, but note the absence of evidence necessary to make an equivalent recommendation for the use of EPT with MSM. Randomized clinical trials to assess the impact of EPT on partner notification, treatment, and STI re-infection among MSM are critical to the development of evidence-based partner management guidelines.

Recent data from urban Peru has identified prevalences of rectal and pharyngeal gonorrhea and chlamydia ranging from 5-20%. The elevated burden of disease among MSM in Peru suggests that frequent transmission of undiagnosed gonorrhea and chlamydia through MSM sexual networks may be a factor contributing to the persistently high incidence of HIV infection among MSM in the region. The investigators propose a pilot evaluation of the effect of EPT on partner notification and treatment among MSM in Peru diagnosed with gonorrhea or chlamydia at any anatomic site.

Specific Aim 1: To explore the social norms and structural factors influencing partner notification and treatment among MSM in Peru.

Specific Aim 2: To determine the effect of EPT on anticipated and actual partner notification among MSM diagnosed with gonorrhea or chlamydia infection.

Specific Aim 3: To develop preliminary data on rates of gonococcal and chlamydial re-infection among MSM randomized to receive EPT compared with standard partner notification counseling.

The proposed study will provide pilot data on the use of EPT with MSM diagnosed with gonorrhea or chlamydia and form the basis for a subsequent Phase III clinical trial of EPT as an STI control method among MSM in Latin America.

DETAILED DESCRIPTION:
Specific Aim 1: To determine the effect of Expedited Partner Therapy (EPT) on anticipated and actual partner notification among MSM diagnosed with gonorrhea or chlamydia infection.

The investigators believe that provision of EPT will alter the behavioral and social contexts of STI management in MSM partnerships by coupling the acts of partner treatment and partner notification. As a result, the investigators hypothesize that MSM provided with EPT will report higher rates of partner notification and treatment compared with men who receive standard partner notification counseling. Quantitative analysis of partner notification outcomes, using the specific examples of participants' five most recent sex partners, will provide a broad estimate of notification and treatment behaviors within the study population. Individual in-depth interviews with a diverse sub-set of participants will be used to provide further interpretive depth regarding the behavioral, social, and structural issues associated with anticipated and actual partner notification and treatment in specific interpersonal contexts, and to address logistical issues related to implementation of the intervention and the accuracy of the study's outcome measures for assessing participants' experiences of partner management.

Specific Aim 2: To collect preliminary data on rates of gonorrhea and chlamydia re-infection among MSM randomized to receive EPT compared with standard partner notification counseling.

The investigators anticipate that MSM provided with EPT will have a lower prevalence of persistent or recurrent urethral, rectal, or pharyngeal gonorrhea and/or chlamydia infection at the one-month follow-up visit compared with men who receive only standard partner notification counseling. Due to the exploratory nature of the proposed study, the investigators have not designed the protocol as an evaluation of the clinical effectiveness of EPT on STI re-infection among MSM. However, the data collected will provide essential preliminary information on the behavioral, social, and epidemiologic contexts of partner management among MSM in Peru needed to design a future clinical trial on the use of EPT as a network-based strategy for STI control among MSM.

Participants will be selected for participation in the study depending on the findings of the EPT/Partner Notification Screening Protocol. Participants in the EPT/Partner Notification Screening Protocol diagnosed with urethritis and/or proctitis, or Gonorrhea and/or Chlamydia in the urethra, rectum, or oropharynx will be eligible for enrollment in the EPT trial protocol.

I. Recruitment: Participants in the EPT/Partner Notification Screening Protocol who are diagnosed by the Study Physician as having clinical urethritis or proctitis, or diagnosed with laboratory-confirmed Gonorrhea and/or Chlamydia infection will be invited by the Study Counselor to participate in the EPT Intervention Protocol.

II. Informed Consent: All potential subjects will receive an explanation of the study procedures and risks and benefits and asked to provide written Informed Consent. Participants will be given the opportunity to take the Informed Consent Document home for further review and decide at a later time if they wish to participate in the study.

III. Enrollment: Subjects who consent to participate in the EPT Intervention Protocol will be randomized to either the Intervention (EPT) or the Standard of Care (Partner Notification Counseling) arm.

IV Randomization: Eligible subjects who provide consent to participate will be randomly assigned to intervention or control groups using a random permuted block allocation (block size=7 in an alternating 4/3 ratio). Computer-generated randomization assignments will be stored in opaque, sealed envelopes opened at the time of allocation. Randomization assignments will be recorded and identified by the participant's numeric study code.

V. Intervention Delivery. Participants assigned to the EPT intervention will be provided with standard partner notification counseling as well as a maximum of 5 EPT packets to distribute to their recent (within 3 months) sex partners.

EPT packets will contain both Cefixime 400 mg and Azithromycin 1g in pill form, as well as a card providing information on gonorrhea and chlamydia infections, the risks and benefits of the antibiotics provided (including allergic reactions), and the importance of testing for HIV and other STIs.

Participants randomized to the control arm will receive standard partner notification counseling by study staff.

Following delivery of the intervention, an appointment will be scheduled for participants to return to the research site in 1 month.

VI. Follow-up Evaluation. All participants will be asked to return to the study site 2-4 weeks after enrollment and randomization. At the Follow-up evaluation, participants will complete a brief survey and undergo repeat testing for gonorrhea/chlamydia.

VII. Survey: Participants will complete a brief follow-up survey assessing the actual notification and treatment outcome for all of their recent partners generally and each of their three most recent partners specifically, as well as factors that impeded and/or promoted partner notification and treatment. Participants will be asked to specify whether each partner was notified, whether they received antibiotic treatment and/or sought HIV/STI testing, the participant's degree of certainty of the outcomes, and the reasons why each partner was or was not notified and/or treated.

VIII. Specimen Collection: Samples of urine, rectal and pharyngeal swabs will be collected as follows:

-Physical Examination: The study physician will conduct a brief physical examination and clinical history to assess for signs or symptoms of STIs, including urethritis, proctitis, and genital ulcer disease. During the physical examination, the study physician will obtain swabs of the rectum and oropharynx. While performing the pharyngeal exam, the physician will use a new Aptima GenProbe collection kit to obtain a swab of the tonsillar pillars. While performing the rectal examination, the physician will use a new Aptima GenProbe collection kit to obtain a swab of the anorectal canal. Participants will also be given the option to self-collect the rectal swab specimen. No urethral swab will be obtained for this study.

Findings from the physical exam and clinical history will be recorded on a Case Report Form (CRF) and identified by the participant's numeric study code.

-Specimen Collection: Following physical examination, participants will be asked to provide a urine sample. Participants will also be instructed in how to collect a 20 mL clean, first-catch urine specimen in a sterile container.

IX. Laboratory Testing: All samples will be tested for the presence of Gonorrhea and Chlamydia at the U.S. Naval Medical Research Unit Laboratory. Participants will be asked to return to the study site in 14 days for results of repeat Gonorrhea and Chlamydia testing. Participants with recurrent or persistent infection will receive a second course of treatment according to the treatment protocol described above. All participants with recurrent or persistent infection will receive additional counseling on the importance of partner notification.

Due to the possibility of fluoroquinolone-resistant gonorrhea infection, participants treated with Ciprofloxacin will be informed of the high frequency of Ciprofloxacin resistance and study staff will emphasize with all participants, but with these participants in particular, the importance of returning to the study site to receive results of their repeat testing/test of cure.

X. Confirmation of Partner Notification: In order to provide independent confirmation of participant-reported notification status, study staff will ask participants for permission to conduct third party partner notification and confirmation of reported notification status. Participants will be asked for permission to contact their recent partner(s) by telephone or e-mail to confirm the notification outcome. Subjects will be informed that they are not obligated to provide contact information for any of their partners. Subjects will also be informed that if they provide contact information for their partner(s), study staff will contact the person using the contact information provided and notify the person only that someone they recently had sex with has been diagnosed with an STI, provide information on local sites offering free or low cost testing for HIV and STIs, and answer any questions the partner might have. Subjects will be informed that study staff will not reveal the participant's name or other identifying information to their partner(s). If the participant provides contact information for their partner(s), study staff will contact the person and provide third-party partner notification using an IRB-approved script. After completing the partner notification process, study staff will ask the partner only if they had previously been notified by a partner about an STI diagnosis ("Yes/No"). Partners will not be asked for any additional information.

XI. Qualitative Evaluation. A randomly selected subgroup of participants in the EPT Intervention Protocol will be invited to participate in individual interviews about the partner notification process. Each participant will be asked to participate in two interviews, one following randomization and one following the Follow-up Visit. Participants will complete a separate informed consent process for the individual interviews and will receive additional compensation for their participation.

XII. Eligibility. A randomly selected subset of participants from the EPT intervention protocol will be invited to participate in the individual qualitative interviews. Every fourth participant randomized will be invited to participate in an individual interview until reaching the projected qualitative study sample of 20 participants (10 each from the intervention and control arms). Participants will be asked to complete a separate informed consent document indicating their willingness to participate in a qualitative interview.

XIII. Interview Conduct. Interviews will be conducted in Spanish in a private room by a trained interviewer. Interviews will be recorded and transcribed verbatim. Participants will be advised that they can stop the interview at any time and that they will be able to stop the tape and erase any response during the interview if they desire.

XIV. Interview Content: Baseline interviews will focus on individual decision-making processes regarding partner notification in specific partnership contexts with a focus on the influence of: STI-related stigma and shame; the gender and sexual identity of participants and their partner(s); perceived power differentials within the partnership(s); patterns of communication within the partnership(s); and structural access to testing and treatment.

Follow-up interviews will discuss actual notification and treatment outcomes. Follow-up interviews will emphasize: barriers or catalysts to implementing notification decisions in specific partnership contexts; the impact of EPT on partner notification practices; practical and logistical issues related to delivery of EPT; structural access to partner testing and treatment within local social, cultural, and economic contexts; and the effectiveness of the study's quantitative outcomes in accurately measuring participants' lived experiences.

Each interview is expected to last approximately 20-30 minutes. Audio recordings and transcripts of interviews will be identified by the participant's numeric study code and the date of the interview.

ELIGIBILITY:
Inclusion Criteria:

1. Biologically male at birth
2. 18 years of age or older
3. Sexual contact (oral or anal intercourse) with a male or male-to-female transgender person within the past 12 months.
4. Clinical Urethritis or proctitis OR Laboratory-diagnosed gonorrhea and/or chlamydia in any anatomic site (urethra, rectum, or oropharynx)

Exclusion Criteria:

1. Under 18 years of age
2. Anatomically female at birth
3. Unable to understand study procedures or provide informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2012-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Self-reported Partner Notification | 21 Days
  Participant self-report of partner notification 14-21 days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Jesse L Clark, MD, MSc, Principal Investigator — University of California, Los Angeles; Thomas J Coates, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Asociacion Civil Impacta Salud y Educacion, Lima, Peru

REFERENCES:
- [Derived] Braun HM, Segura ER, Lake JE, Gandhi M, Rios J, Villaran MV, Sanchez J, Lama JR, Clark JL. Individual and partnership factors associated with anticipated versus actual partner notification following STI diagnosis among men who have sex with men and/or with transgender women in Lima, Peru. Sex Transm Infect. 2018 Dec;94(8):607-610. doi: 10.1136/sextrans-2017-053292. Epub 2017 Nov 30. PMID 29191814
- [Derived] Clark JL, Segura ER, Oldenburg CE, Rios J, Montano SM, Perez-Brumer A, Villaran M, Sanchez J, Coates TJ, Lama JR. Expedited Partner Therapy (EPT) increases the frequency of partner notification among MSM in Lima, Peru: a pilot randomized controlled trial. BMC Med. 2017 May 4;15(1):94. doi: 10.1186/s12916-017-0858-9. PMID 28468648